CLINICAL TRIAL: NCT05246748
Title: Does Watson's Human Caring Theory-based Breastfeeding Educational and Support Programme Affects Mothers Breastfeeding Self-efficacy, Duration, Definitions and Satisfaction?: A Randomised Controlled Trial
Brief Title: Human Caring Theory-based Breastfeeding Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gamze Durmazoğlu (Other)
Responsible Party: Sponsor-Investigator, Gamze Durmazoğlu, Principal Investigator, Dokuz Eylul University
Organization: Dokuz Eylul University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GmZ!2805
Record Dates: First submitted 2022-01-21; First posted 2022-02-18 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: Breastfeeding Education
Keywords: Theory of Human Caring; Breastfeeding; Nursing; Self-efficacy
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group was given a breastfeeding education program based on the HCT for six face to face sessionconducted in parallel with asynchronous distance education sessions in prenatal period and continued with web based sessions and telephone support in postnatal period.
  Interventions: Other: Human Caring Theory based Education
- Control group (Active Comparator): The control group received solely standard education program for one sessions in prenatal period.
  Interventions: Other: Standard Education

INTERVENTIONS:
Other: Human Caring Theory based Education — The intervention group was given a breastfeeding education program based on the HCT for six face to face sessionconducted in parallel with asynchronous distance education sessions in prenatal period and continued with web based sessions and telephone support in postnatal period.
  Arms: Intervention group
Other: Standard Education — The control group received solely standard education program for one sessions in prenatal period.
  Arms: Control group

SUMMARY:
It is a randomized controlled prospective study. The purpose of the study is to examine the effect of breastfeeding education and support program based on Human Caring Theory (HCT) on mothers' breastfeeding self-efficacy, duration and definitions, and their satisfaction with this process. As a result, Human Caring Theory based breastfeeding education program improved breastfeeding self-efficacy, duration and exclusive breastfeeding.

DETAILED DESCRIPTION:
Although breastfeeding have many benefits, breastfeeding rates are still not at the desired level. One of the most important factors in increasing breastfeeding rates is breastfeeding education. Therefore, the purpose of the study is to examine the effect of breastfeeding education and support program based on Human Caring Theory (HCT) on mothers' breastfeeding self-efficacy, duration and definitions, and their satisfaction with this process.

It is a randomized controlled prospective study conducted between January 2019- March 2020 in 100 Turkish women (intervention:50; control: 50). A simple randomization method was performed using the siterandomizer.org to ensure samples' equality in two groups. The participants were randomly assigned to the groupwith Human Caring Theory based education and support (intervention) or a standard education program (control) group. The study method was explained, and informed consent was obtained from all participants. The researcher applied the education and support, and hence, blinding could not be done.

An intervention program was prepared by researchers who received many trainings on the practical use of Watson Human Caring theory. Watson Human Caring Theory based education and support program was conducted in groups of 6-8 pregnant woman in prenatal period and continues individualty web- based and by phone support in postnatal period. Two experts who have PhD degree in women's health nursing assessed the validity of the breastfeeding education program based on the HCT. The intervention group was given a breastfeeding education program based on the HCT for six face to face session conducted in parallel with asynchronous distance education sessions in prenatal period and continued with web based sessions and telephone support in postnatal period. The control group received solely standard education program for one sessions in prenatal period. Especially in postnatal period traditional face-to-face breastfeeding education and support may not be easy for women and their families. The "Breastfeeding Self-Efficacy Scale", "Baby's Feeding Definition Form" and "Watson Caritas Patient Score"instruments were used for data collection.

Women's Descriptive Characteristics Question Form, The Baby's FeedingDefinition Form, Breastfeeding Self- Efficacy Scale-Short Form and Watson Caritas Patient Score were the instruments used for data collection.

Women's Descriptive Characteristics Question Formincluded ten questions related to age, education level, previous breastfeeding educationand gestational age.

In order to asses baby's feeding, The Baby Feeding Definition Form was used. This form was prepared by researchers in line with literatüre. The questions such as the baby's sucking status, the status of receiving liquid or nutrients other than breast milk, and the baby's appearance of peace after sucking were based on Labbok and Krasovec (1990) and WHO classificationts relted to baby breast milk intake level. At the same time the state of peace of the baby was evaluated according to the expressions of the mothers. Consequently three breastfeeding experts evaluated the form and found it suitable for the assessment of infants' feeding level. The responses obtained from the evaluation form were classified according to the diagnostic criteria for breastfeeding by Labbok and Krosovec (1990).

The Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF) comprised 14 items developed by Dennis in 2003. The BSES-SFis a 5-point Likert-type scale, with 1meaning "not at all confident" and 5 meaning "very confi-dent," yielding a minimum possible score of 14 points and a maximum score of 70 points. Regarding this scale a high score indicates high breast-feedingself-efficacy. The scale had a Cronbach's alpha value of 0.94. Turkish validity and reliability of the scale were done by Tokat, Okumuş and Dennis (2010). In the same study, Cronbach's alpha coefficient for internal consistency was 0.87 antenatally and 0.86 postnatally. Prenatal items was created by using the future tense expression in the antenatal form of the breastfeeding self-efficacy scale.

The Watson Caritas Patient Score (WCPS) was used to assess satisfaction of the education program. WCPS was developed based on caritas factors and caritas processes by Dr. Jean Watson et al. (2010). WCPS is a reliable and valid instrument used in hospitals and systems to assess perspectives of caring practices of hospital staff, of colleagues and peers.The WCPS items are each scored on a 7-point scale, ranging from "not at all" (1) to "very much" (7). The reliability was confirmed with a Cronbach's α of .90. (Brewer & Watson, 2015). The internal consistency of the WCPS assessed using Cronbach's alpha was .90 in Turkey (Durmazoglu, 2020).The highest score that can be obtained from WCPS is 35, and the lowest score is five. In this form there is also comments and suggestions section. In this section people can write their comments for more effective process.

The data were analyzed using the Statistical Package for Social Sciences (SPSS 22.0) for Windows. The normal distribution of the data was evaluated using the Kolmogorov-Smirnov test. The descriptive statistics of the study were evaluated with frequency, mean, standard deviation, number and percentage. Pearson's chi-square test was used to evaluate the homogeneity of the data according to the groups. The t-test was used for comparisons between variables in two categories. Multiple and one-way analysis of variance was used for repeated measurements. The reliability of the scales was tested with Cronbach's alpha. The significance threshold was set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous women with 28-34 weeks of pregnancy able to speak and understand Turkish without any communication barrier were

Exclusion Criteria:

* Having some (a) maternal problems (mastectomy, mastitis and drug use, psychiatric diseases, etc.),or (b) infant problems(cleft palate, chromosomal anomalies, neurological diseases that will adversely affect breastfeeding, etc.) were determined as exclusion criteria.

Ages: 19 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
BREASTFEEDİNG SELF-EFFİCACY | Change from breastfeeding self-efficacy at 6 months
  BREASTFEEDİNG SELF-EFFİCACY SCORE
BREASTFEEDİNG DURATION | Change from breastfeeding duration at 6 months
  HOW LONG BREASTFEEDİNG CONTİNUES
THE BABY FEEDİNG DEFİNİTİON FORM | Change from the babies breastfeeding definition at 6 months
  EXPLAINS THE TYPE OF BREASTFEEDING.SUCH AS EXCLUSİVE BREASTFEEDİNG OR PARİTAL BREASTFEEDİNG ETC.
WATSON CARİTAS PATİENT SCORE | 1 week
  DETERMINES WOMEN'S SATISFACTION LEVELS WITH THE EDUCATION THEY RECEIVE. IN THIS STUDY, MOTHERS WITH HIGH WATSON CARITAS PATIENT SCORES ALSO HAVE HIGH LEVELS OF SATISFACTION WITH THE EDUCATION PROCESS.

CONTACTS AND LOCATIONS:
Locations (1):
- Gamze DURMAZOĞLU, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Starting after publication
Access Criteria: Researchers who study for women and child health can review requests and criteria for reviewing requests may also be provided.

REFERENCES:
- [Background] Almohanna AA, Win KT, Meedya S. Effectiveness of Internet-Based Electronic Technology Interventions on Breastfeeding Outcomes: Systematic Review. J Med Internet Res. 2020 May 29;22(5):e17361. doi: 10.2196/17361. PMID 32469315
- [Background] Alus Tokat M, Okumus H, Dennis CL. Translation and psychometric assessment of the Breast-feeding Self-Efficacy Scale-Short Form among pregnant and postnatal women in Turkey. Midwifery. 2010 Feb;26(1):101-8. doi: 10.1016/j.midw.2008.04.002. Epub 2008 Jun 9. PMID 18541350
- [Background] Arslan-Ozkan I, Okumus H, Buldukoglu K. A randomized controlled trial of the effects of nursing care based on Watson's Theory of Human Caring on distress, self-efficacy and adjustment in infertile women. J Adv Nurs. 2014 Aug;70(8):1801-12. doi: 10.1111/jan.12338. Epub 2013 Dec 22. PMID 24372443
- [Background] Bai YK, Lee S, Overgaard K. Critical Review of Theory Use in Breastfeeding Interventions. J Hum Lact. 2019 Aug;35(3):478-500. doi: 10.1177/0890334419850822. Epub 2019 May 17. PMID 31100027
- [Background] Bensley RJ, Hovis A, Horton KD, Loyo JJ, Bensley KM, Phillips D, Desmangles C. Accessibility and preferred use of online Web applications among WIC participants with Internet access. J Nutr Educ Behav. 2014 May-Jun;46(3 Suppl):S87-92. doi: 10.1016/j.jneb.2014.02.007. PMID 24810002
- [Background] Boateng GO, Martin SL, Tuthill EL, Collins SM, Dennis CL, Natamba BK, Young SL. Adaptation and psychometric evaluation of the breastfeeding self-efficacy scale to assess exclusive breastfeeding. BMC Pregnancy Childbirth. 2019 Feb 18;19(1):73. doi: 10.1186/s12884-019-2217-7. PMID 30777020
- [Background] Brewer BB, Watson J. Evaluation of Authentic Human Caring Professional Practices. J Nurs Adm. 2015 Dec;45(12):622-7. doi: 10.1097/NNA.0000000000000275. PMID 26502069
- [Background] Brockway M, Benzies K, Hayden KA. Interventions to Improve Breastfeeding Self-Efficacy and Resultant Breastfeeding Rates: A Systematic Review and Meta-Analysis. J Hum Lact. 2017 Aug;33(3):486-499. doi: 10.1177/0890334417707957. Epub 2017 Jun 23. PMID 28644764
- [Background] Cangöl, E., Hotun Şahin, N. (2017). A Model of Breastfeeding Support: Motivational Interviews Based On Pender's Health Promotion Model. HJournal of Education and Research in Nursing, 14 (1), 98-103. doi: 10.5222/HEAD.2017.098
- [Background] Chan MY, Ip WY, Choi KC. The effect of a self-efficacy-based educational programme on maternal breast feeding self-efficacy, breast feeding duration and exclusive breast feeding rates: A longitudinal study. Midwifery. 2016 May;36:92-8. doi: 10.1016/j.midw.2016.03.003. Epub 2016 Mar 8. PMID 27106949
- [Background] Chauhan SP, Blackwell SC, Saade GR; Society for Maternal-Fetal Medicine Health Policy Committee. A suggested approach for implementing CONSORT guidelines specific to obstetric research. Obstet Gynecol. 2013 Nov;122(5):952-956. doi: 10.1097/AOG.0b013e3182a9c9af. PMID 24104788
- [Background] Chipojola R, Chiu HY, Huda MH, Lin YM, Kuo SY. Effectiveness of theory-based educational interventions on breastfeeding self-efficacy and exclusive breastfeeding: A systematic review and meta-analysis. Int J Nurs Stud. 2020 Sep;109:103675. doi: 10.1016/j.ijnurstu.2020.103675. Epub 2020 Jun 6. PMID 32585447
- [Background] Dennis CL. Identifying predictors of breastfeeding self-efficacy in the immediate postpartum period. Res Nurs Health. 2006 Aug;29(4):256-68. doi: 10.1002/nur.20140. PMID 16847899
- [Background] Dennis CL. The breastfeeding self-efficacy scale: psychometric assessment of the short form. J Obstet Gynecol Neonatal Nurs. 2003 Nov-Dec;32(6):734-44. doi: 10.1177/0884217503258459. PMID 14649593
- [Background] Dennis CL. Theoretical underpinnings of breastfeeding confidence: a self-efficacy framework. J Hum Lact. 1999 Sep;15(3):195-201. doi: 10.1177/089033449901500303. No abstract available. PMID 10578797
- [Background] Diji AK, Bam V, Asante E, Lomotey AY, Yeboah S, Owusu HA. Challenges and predictors of exclusive breastfeeding among mothers attending the child welfare clinic at a regional hospital in Ghana: a descriptive cross-sectional study. Int Breastfeed J. 2017 Mar 9;12:13. doi: 10.1186/s13006-017-0104-2. eCollection 2016. PMID 28286540
- [Background] Durmazoglu G, Yenal K, Okumus H. Maternal Emotions and Experiences of Mothers Who Had Breastfeeding Problems: A Qualitative Study. Res Theory Nurs Pract. 2020 Jan 1;34(1):3-20. doi: 10.1891/1541-6577.34.1.3. PMID 31937633
- [Background] Finfgeld-Connett D. Meta-synthesis of caring in nursing. J Clin Nurs. 2008 Jan;17(2):196-204. doi: 10.1111/j.1365-2702.2006.01824.x. Epub 2007 Mar 1. PMID 17331089
- [Background] Gu Y, Zhu Y, Zhang Z, Wan H. Effectiveness of a theory-based breastfeeding promotion intervention on exclusive breastfeeding in China: A randomised controlled trial. Midwifery. 2016 Nov;42:93-99. doi: 10.1016/j.midw.2016.09.010. Epub 2016 Sep 22. PMID 27788416
- [Background] Khorshidifard, M., Amini, M., Dehghani, M.R., Zaree, N., et al. (2017). Assessment of breastfeeding education by face to face and small-group education methods in mothers' self-efficacy in Kazeroun Health Centers in 2015. Women's Health Bulletin, 4(3), 2-6.doi: 10.5812/WHB.41919
- [Background] Kim SK, Park S, Oh J, Kim J, Ahn S. Interventions promoting exclusive breastfeeding up to six months after birth: A systematic review and meta-analysis of randomized controlled trials. Int J Nurs Stud. 2018 Apr;80:94-105. doi: 10.1016/j.ijnurstu.2018.01.004. Epub 2018 Jan 12. PMID 29407349
- [Background] Koskinen KS, Aho AL, Hannula L, Kaunonen M. Maternity hospital practices and breast feeding self-efficacy in Finnish primiparous and multiparous women during the immediate postpartum period. Midwifery. 2014 Apr;30(4):464-70. doi: 10.1016/j.midw.2013.05.003. Epub 2013 Jun 13. PMID 23768951
- [Background] Labbok M, Krasovec K. Toward consistency in breastfeeding definitions. Stud Fam Plann. 1990 Jul-Aug;21(4):226-30. PMID 2219227
- [Background] Lau CYK, Lok KYW, Tarrant M. Breastfeeding Duration and the Theory of Planned Behavior and Breastfeeding Self-Efficacy Framework: A Systematic Review of Observational Studies. Matern Child Health J. 2018 Mar;22(3):327-342. doi: 10.1007/s10995-018-2453-x. PMID 29427014
- [Background] Lewkowitz AK, Cahill AG. Mobile Health Approaches to Breastfeeding. Clin Obstet Gynecol. 2021 Jun 1;64(2):384-391. doi: 10.1097/GRF.0000000000000606. PMID 33813523
- [Background] Loke AY, Chan LK. Maternal breastfeeding self-efficacy and the breastfeeding behaviors of newborns in the practice of exclusive breastfeeding. J Obstet Gynecol Neonatal Nurs. 2013 Nov-Dec;42(6):672-84. doi: 10.1111/1552-6909.12250. Epub 2013 Oct 15. PMID 24128113
- [Background] Ozan, Y.D., Okumuş, H. (2013). Nursing Care of Women with Unsuccessful Infertility Treatment According to Watson's Theory of Caring. Anatolian Journal of Nursing and Health Sciences, 16, 3.
- [Background] Özkara, H., Fidancı, B.E., Yıldız, D., Kaymakamgil, Ç. (2016). Lactation consult. TAF Preventive Medicine Bulletin, 15(6), 551- 555. doi: 10.5455/pmb.1-1436701913
- [Background] Parry KC, Tully KP, Hopper LN, Schildkamp PE, Labbok MH. Evaluation of Ready, Set, BABY: A prenatal breastfeeding education and counseling approach. Birth. 2019 Mar;46(1):113-120. doi: 10.1111/birt.12393. Epub 2018 Sep 6. PMID 30191591
- [Background] Şengün, F., Üstün, B., & Bademli, K. (2013). Exploration of Theory/Model Based Nursıng Research In Turkey. Anatolian Journal of Nursing and Health Sciences, 16(2), 132-139.
- [Background] Tokat, M.A., & Okumus, H. (2013). Mothers Breastfeeding Self-Efficacy and Success: Analysis The Effect of Education Based on Improving Breastfeeding Self-Efficacy. Journal of Education and Research in Nursing, 10(1), 21-29.
- [Background] Tseng JF, Chen SR, Au HK, Chipojola R, Lee GT, Lee PH, Shyu ML, Kuo SY. Effectiveness of an integrated breastfeeding education program to improve self-efficacy and exclusive breastfeeding rate: A single-blind, randomised controlled study. Int J Nurs Stud. 2020 Nov;111:103770. doi: 10.1016/j.ijnurstu.2020.103770. Epub 2020 Sep 3. PMID 32961461
- [Background] van Dellen SA, Wisse B, Mobach MP, Dijkstra A. The effect of a breastfeeding support programme on breastfeeding duration and exclusivity: a quasi-experiment. BMC Public Health. 2019 Jul 24;19(1):993. doi: 10.1186/s12889-019-7331-y. PMID 31340787
- [Background] Watson, J., Brewer, B.B., D'Alfonso, J. (2010). Watson caritas patient score (WCPS). Watson Caring Science Institute: Boulder, CO. Accessed: www.watsoncaringscience.org Last accessed: 27.11.2021
- See also: Global Nutrition Targets 2025 Breastfeeding Policy Brief — https://apps.who.int/iris/handle/10665/149022